CLINICAL TRIAL: NCT00376870
Title: Prevention of Coronary Artery in STENT Restenosis With the Combined Use of Pioglitazone and Sirolimus-Eluting Coronary Stent
Brief Title: PIoglitazone for PrEvention of Restenosis in Diabetic Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Fabrizio Clementi, Fabrizio Clementi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PIPER
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2008-08-01 (Estimated); Status verified 2008-06

CONDITIONS: Coronary Atherosclerosis; Coronary Restenosis; Diabetes
Keywords: PCI; STENT; Coronary; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis; Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone (Active Comparator): Pioglitazone 30mg/d
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — pioglitazone 30 mg/d
  Arms: Pioglitazone
Drug: Placebo — Placebo 30 mg/d
  Arms: Placebo

SUMMARY:
Restenosis requiring reintervention is still a limitation of percutaneous coronary angioplasty. Despite the use of Drug eluting stent (DES), the rate of restenosis remains 7% to 16% in diabetic patients, making it a challenging problem in interventional cardiology.

Still, in clinical trials, most of these attempts did not successfully limit neointimal formation after coronary stenting.

Thiazolidinediones (TZDs), like pioglitazone (pio) or rosiglitazone, are a novel class of oral antidiabetic agents currently used to treat patients with type 2 diabetes mellitus.

These agents increase insulin sensitivity and, as such, have favorable effects on blood glucose levels and the lipid profile in treated patients.

Beyond their metabolic action, TZDs have been shown to exhibit antiinflammatory and antiatherogenic effects in vascular cells in vitro and to limit lesion development in various animal models of arteriosclerosis.

Moreover, TZDs inhibit VSMC proliferation and migration, 2 critical processes in neointimal formation after coronary stenting.

Data from rodent models suggest that TZDs limit intimal proliferation after vascular injury, and in clinical studies with type 2 diabetic coronary artery disease (CAD) patients, TZDs have been shown to reduce neointimal formation as well as restenosis after coronary stent implantation.

Still, it remains unclear to what extend these effects depend on the metabolic action of these drugs and what might mainly be due to the improvement in glycemic control.

Recently a few reports on prevention of restenosis in type 2 diabetic patients (T2DM) with the use of TZDs as been published. All of them uses BMS as endoprosthetic devices. None of these evaluated the use of TZDs in combination with DES.

Aim of the study is to evaluate the efficacy of pioglitazone in prevention of in-stent restenosis after successful implantation of a sirolimus-eluting coronary stent for treatment of de-novo "complex" coronary vessel disease in patients with T2DM and stable coronary artery disease.

Study primary end-point are late-loss at 9 months.Secondary end-point include binary restenosis MACE at 1, 9 and 12 month, stent thrombosis at 12 months.

DETAILED DESCRIPTION:
2.Design This is a randomised, placebo-controlled, double-blinded, multicenter centre study.The patients' clinical data will be recorded on case report forms (CRF).

3.Aim of the study To evaluate the efficacy of Pioglitazone (30 mg/daily) therapy on in-stent late luminal loss in T2DM patients treated with sirolimus-eluting stent for a complex lesion. Both Pioglitazone and matched Placebo will be provided by Takeda Global Research & Development (TGRD), London, UK.

4.Endpoints

4.1.Primary Endpoint

The primary end-point is defined by:

* In-stent late luminal loss after 9 months of implant procedure

4.2.Secondary Endpoint

The secondary end-points are defined by:

* Binary restenosis (defined as in-segment stenosis of at least 50 percent on follow-up angiography)
* Incidence of major adverse cardiac events (MACE) within discharge, 30 days, 6 and 12 months after implant procedure. The major adverse events are described as follows:

  * Acute myocardial infarction
  * Cardiac death;
  * Recurrent Myocardial infarction (Q-wave and non-Q wave)
  * Target Lesion Revascularization (TLR)
  * Target Vessel Revascularization (TVR)
* Incidence of STENT Thrombosis classified by the ARC definition:

  * definite, probable, or possible
  * Acute (0 to 24 hours after stent implantation), Subacute ( >24 hours to 30 days), or Late (>30 to 360 days) and Very Late (> 1 year afer stent implantation).
* Safety and tolerability

  5.Study population Sample size is calculated on the basis of results from previous trials that have examined the effect of TZDs on neointima formation in diabetic subjects, with late luminal loss in the control group of 0.43±0.45 mm and a pre-specified 40% reduction in the TZDs group (expected late luminal loss of 0.26±0.28 mm) resulting in 86 lesions per group to achieve statistical significance ([alpha]=0.05, [beta]=0.2, 2 tailed). Considering a 20% of patients lost in follow-up and a mean of 1.3 lesion for patients treated we will need 80 patients per group. The patients to be enrolled have to fulfil the inclusion criteria listed below and none of the exclusion criteria and they have to be enrolled in a consecutive manner.

  6.Conduct of the study

6.1.Screening procedure and enrollment Patients with T2DM, scheduled for angioplasty will be screened for eligibility. If all inclusion criteria are met and no exclusion criteria are present the patients should be enrolled in the study.

6.2 Randomisation procedure After informed written consent is obtained a randomisation number will be assigned to the patient. A pre-packed blind-label study drug or placebo with a 3 months dose will be assigned to the patient. The first dose will be administered before the implant procedure and continued for 9 months. Randomisation code will be stored in a safe place.

6.3 Stenting procedure Stents can be implanted after lesion predilatation, or using direct stenting technique, performed at the discretion of the operator. After checking the correct position, stent should be inflated and deployed with a single inflation. Residual stenosis, after the stent implant, must be less than 10%. If needed another stent should be placed overlapping with former. Post dilatation of the overlapped segment, with a non-compliant balloon is mandatory.

6.4 Pharmacological treatment

Pre-procedure:

* Aspirin 75 mg
* Clopidogrel loading dose of 600 mg

Intravenous GP IIb/IIIa agents will be allowed at the discretion of the operator with the following doses:

* Abciximab 0,25 mg/kg intravenous bolus 10-60 min. before the procedure, followed by a continuous infusion of 0,125 mg/kg/min for 12-18 hours.
* Tirofiban 10 mcg/kg intravenous bolus, followed by a continuous infusion of 0, 15 mcg/kg/min for 18-24 hours.
* Eptifibatide 180 mcg/kg intravenous bolus immediately before the procedure, followed by a continuous infusion of 2 mcg/kg/min (in patients with serum creatinine > 2 mg/dl the infusion should be of 1 mcg/kg/min) and a second bolus of 180 mcg/kg/min 10 min. after the first bolus. Infusion should be maintained for 18-24 hours.

Intra-procedure:

*Heparin will be given at the dose of 70-100 U/kg if no GP IIb/IIIa are administered or at a dose of 50/70 U/Kg if GP IIb/IIIa are administered.

Post-procedure:

*Aspirin 75 mg/day indefinitely

*Clopidogrel 75 mg/day for 12 months All of the patients will receive standard medical therapy as judged by the reference cardiologist, including, [beta]-blockers, angiotensin-converting enzyme inhibitors, and statins.

7.In hospital and follow-up examination

Physical examination:

A physical examination will be performed in all patients enrolled before hospital discharge, and at 3, 9 and 12 months. The physical evaluation must include an assessment of the patient's clinical status, including evaluation of ischemia and angina status.

The patient and primary care physicians will be strongly encouraged to keep an "optimal" control of the glycemia, considering the following recommendation:

Changes in life style with increment in physical activity will be suggested for all patients. The diabetology centre will treat patients with stepwise approach to achieve a possible goal of HbA1c < 7% and daily glycaemic levels reported in the following table.

Glycemic goals ADA and AACE criteria (1,2) HbA1c 6.5 - 7.0% Fasting / pre-prandial glucose levels 90 - 130 mg/dl Post-prandial glucose levels 140 - 180 mg/dl Bed time glucose levels 110 - 150 mg/dl

1. American Diabetes Association, Diabetes Care 2004, 27: S15-S35
2. American Association of Clinical Endocrinologists, Endocrine Pract 2002 (suppl.1): 40-82.

The approach will be:

* Type 2 diabetic patients on oral anti-diabetic (OAD) therapy

  1. starting with OAD monotherapy,
  2. if failure after 2 months (HbA1c>7.0%), OAD monotherapy uptitration
  3. if failure (HbA1c>7.0%), OAD combination
  4. if failure (HbA1c>7.0%), OAD + basal insulin
  5. if failure (HbA1c>7.0%), OAD + multiple daily insulin injections
  6. if failure (HbA1c>7.0%), multiple daily insulin injections Starting from point 3, diabetology centre will decide on the dosing and therapeutic regimens. Type 2 diabetic patients on insulin therapy
  7. Multiple daily insulin injections, with increasing doses if HbA1c>7.0% The number of diabetologic follow-up visits will be decided by the usual diabetology care policy of the centre according to plasma glucose and HbA1c levels

     Blood samples: cardiac enzymes (Troponin, CK and CK-MB) should be evaluated before the procedure and before discharge (CK-MB after 6, 12 and 24 hour and continued if abnormal till normalization).

     Metabolic and inflammatory indices will be analysed before discharge and at 3, 9 and 12 months follow-up. Among them will be evaluated: fasting glucose, fasting insulin, HbA1c, triglyceride, total cholesterol, LDL cholesterol, HDL cholesterol, APO-a/APO-b, Hs-CRP, CD40L, Adiponectin.
  8. Scheduled follow-up visit

     Patients will be contacted by phone at 30 days and 6 months follow-up and they will undergo clinical evaluation after 3, 9 and 12 months. At 9 months follow-up, patients will be scheduled for a repeat angiography.

     Pre procedure Post procedure Hospital discharge 30-day follow-up 3 month follow-up 6 month follow-up 9 month follow-up 12 month follow-up Physical examination Yes - Yes Phone call Yes Phone call Yes Yes Blood sampling Yes Ck-MB, CK, Tn - - Yes Yes Yes Coronary angiography Yes Yes - - - Yes -
  9. Definitions

9.1 In segment late-luminal loss

Defined as difference between the minimal luminal diameter at the end of the procedure and the minimal luminal diameter at 9 months follow-up in the target lesion or either edge (5mm).

9.2 Major Adverse Cardiac Events

Acute Myocardial infarction: Chest pain persisting for > 30 minutes associated with:

ST segment elevation of at least 0.1 mV in two or more contiguous leads; or true posterior MI with ST segment depression of at least 0.1 mV in leads V1 through V3; or new left bundle branch block; and elevation of CK-MB or CK more than two times upper limit of normal. Periprocedural myocardial infarction is defind by > 3 times ULN rise in troponin or CK-MB

Cardiac death: all deaths occurring during the study are considered cardiac related unless clinical assessment can establish an unequivocal non-cardiac cause.

Re-infarction: a diagnosis of a new myocardial infarction is clinically defined on the basis of ECG or enzymatic doses if one of the following criteria is met:

1. Detection of new pathological Q-waves not present on baseline ECG according to the Minnesota Code.
2. Enzyme changes defined by more than two times upper limit of normal CK and the presence of CK-MB. If the CK-MB is not available, the CK will be accepted as evidence of myocardial infarction.

Target lesion revascularization: repeat revascularization (PCI or CABG) in the follow-up period due to restenosis either in the target lesion or either edge (5mm).

Target vessel revascularization: repeat revascularization (PCI or CABG) in the follow-up period due to restenosis either within the target lesion or anywhere else in the same epicardial coronary artery (includes proximal and distal lesions, branches and left main).

9.3 Binary restenosis

Defined as in-segment stenosis of at least 50 percent on follow-up angiography.

9.4 Thrombosis

The definition of definite stent thrombosis required the presence of an acute coronary syndrome with angiographic or autopsy evidence of thrombus or occlusion.

Probable stent thrombosis included unexplained deaths within 30 days after the procedure or acute myocardial infarction involving the target-vessel territory without angiographic confirmation.

Possible stent thrombosis included all unexplained deaths occurring 30 days after the procedure.

9.5 Complex Lesion definition

* Total occlusions.
* Long lesions (≥ 28 mm). Two long lesions in series necessitating overlapping stents are accepted.
* True bifurcation lesions with a side branch greater than or expected to be ≥2.5 mm by visual estimate.
* Patients requiring 4 or more stents in one procedure.
* Target lesions in a vessels with diameter 2.5 mm by visual estimate which are not secondary branches such as postero-laterals, diagonals or obtuse marginals.

  10. Quantitative Coronary Angiography Baseline, postprocedural, and follow-up coronary angiograms will be digitally recorded and assessed off-line in the angiographic laboratory with an automated edge-detection system by experienced personnel unaware of the study drug allocation. The complexity of the lesions will defined according to the modified grading system of the American College of Cardiology-American Heart Association16 . The morphologic appearance of in-stent restenosis at follow-up angiography will be classified according to the system proposed by Mehran et al.17. All measurements will be performed on cineangiograms recorded after the intracoronary administration of nitroglycerin. The same single, worst-view projection will be used at all times. The contrast-filled nontapered catheter tip will be used for calibration. The reference diameter will be determined by interpolation.

The variables that will be measured include the reference diameter of the vessel, the minimal diameter of the lumen, the extent of stenosis (the difference between the reference diameter and the minimal luminal diameter, divided by the reference diameter and multiplied by 100), late luminal loss (the difference between the minimal luminal diameter at the end of the procedure and the minimal luminal diameter at 9 follow-up), and net luminal gain (the difference between the minimal luminal diameter at 9 follow-up and the minimal luminal diameter before the procedure). Quantitative analysis will be used to evaluate the stented area ("in stent") and the area that included the stented segment as well as the 5-mm margins proximal and distal to the stent ("in segment").

12. Safety and Tolerability

12.1 Definition of Adverse Events (AE) An AE is defined as any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product; it does not necessarily have to have a causal relationship with this treatment.

An AE can therefore be any unfavourable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not it is considered related to the medicinal product.

12.2 Definition of Serious Adverse Events (SAE)

A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose:

1. Results in DEATH.
2. Is LIFE THREATENING.

   • The term "life threatening" refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it were more severe.
3. Requires inpatient HOSPITALIZATION or prolongation of existing hospitalization.
4. Results in persistent or significant DISABILITY/INCAPACITY.
5. Leads to a CONGENITAL ANOMALY/BIRTH DEFECT.
6. Is an IMPORTANT MEDICAL EVENT that satisfies any of the following:

   * May require intervention to prevent items 1 through 5 above.
   * May expose the subject to danger, even though the event is not immediately life threatening or fatal or does not result in hospitalization.
   * Includes any event or synonym described in the Takeda Medically Significant List (Table A):

Table A Takeda Medically Significant List Term Acute respiratory failure/acute respiratory distress syndrome Hepatic necrosis Ventricular fibrillation Acute liver failure Torsade de pointes Anaphylactic shock Malignant hypertension Acute renal failure Convulsive seizures Pulmonary hypertension Agranulocytosis Pulmonary fibrosis Aplastic anemia Confirmed or suspected endotoxin shock Toxic epidermal necrolysis Confirmed or suspected transmission of infectious agent by products Stevens-Johnson syndrome

12.3 Severity of AEs

The different categories of intensity (severity) are characterized as follows:

Mild: The event is transient and easily tolerated by the subject. Moderate: The event causes the subject discomfort and interrupts the subject's usual activities.

Severe: The event causes considerable interference with the subject's usual activities.

12.4 Causality of AEs

The relationship of each AE to study drug will be assessed using the following categories:

Definite: An AE that follows a reasonable temporal sequence from administration of the drug (including the course after treatment withdrawal of the drug) AND that satisfies any of the following:

* Reappearance of similar reaction upon readministration (rechallenge).
* Positive results in a drug sensitivity test (skin test, etc).
* Toxic level of the drug revealed by measurement of drug concentrations in blood or another body fluid.

Probable: An AE that follows a reasonable temporal sequence from administration of the drug (including the course after withdrawal of the drug) AND for which involvement of factors other than the drug, such as underlying diseases, complications, concomitant drugs, and concurrent treatment can reasonably be excluded.

Possible: An AE that follows a reasonable temporal sequence from administration of the drug (including the course after withdrawal of the drug) AND for which possible involvement of the drug can be argued although factors other than the drug, such as underlying diseases, complications, concomitant drugs, and concurrent treatments also may be responsible. For example, there have been similar reports in the past, including reports on its analogues, or the occurrence of the event could be predicted from the pharmacologic actions or chemical structure of the drug.

Not related: An AE that does not follow a reasonable temporal sequence from administration of the drug or that can be reasonably explained by other factors, such as underlying diseases, complications, concomitant drugs, and concurrent treatments.

12.5 Relationship to Study Procedures

Relationship (causality) to study procedures should be determined for AEs. The relationship should be assessed as "Yes" if the investigator considers that there is reasonable possibility that an event is due to a study procedures. Otherwise, the relationship should be assessed as "No".

12.6 AE Reporting

At each study visit, the investigator will assess whether any subjective AEs have occurred. A neutral question, such as "How have you been feeling since your last visit?" may be asked. Subjects may report AEs occurring at any other time during the study.

All subjects experiencing AEs, whether considered associated with the use of the study medication or not, must be monitored until the symptoms subside and any clinically relevant changes in laboratory values have returned to baseline or until there is a satisfactory explanation for the changes observed. All AEs will be documented in the AE page of the CRF, whether or not the investigator concludes that the event is related to the drug treatment. The following information will be documented for each event:

* Event term.
* Start and stop date and time.
* Severity.
* Investigator's opinion of the causal relationship between the event and administration of study drug(s) (not related, possible, probable, or definite).
* Investigator's opinion of the causal relationship to study procedure(s), including the details of the suspected procedure.
* Action concerning study drug.
* Outcome of event.

12.7 Collection and Reporting of SAEs

When an SAE occurs after informed consent through the AE collection period it should be reported according to the following procedure:

A Takeda SAE form must be completed, in English, and signed by the investigator immediately or within 1 working day of first onset or notification of the event. The information should be completed as fully as possible but contain, at a minimum:

* A short description of the event and the reason why the event is categorized as serious.
* Subject identification number.
* Investigator's name.
* Causality assessment.

The SAE form should be transmitted within 1 working day to the attention of:

Takeda Global Research & Development (TGRD) Pharmacovigilance Dept. Arundel Great Court, 2 Arundel Street London WC2R 3DA Fax No: + 44 207 759 5272

Any SAE spontaneously reported to the investigator following the AE collection period should be reported to TGRD.

12.8 Follow-up of SAEs

If information not available at the time of the first report becomes available at a later date, the investigator should add this to the initial SAE form or provide other written documentation and fax it immediately within 1 working day of receipt. Copies of any relevant data from the hospital notes (eg, ECGs, laboratory tests, discharge summary, postmortem results) should be sent to the addressee, if requested.

All SAEs should be followed up until resolution or permanent outcome of the event. The timelines and procedure for follow-up reports are the same as those for the initial report.

13. Patient withdrawal

Patient may withdraw from the study at any time and for any reason, without affecting their right to treatment by the Investigator. Every patient should be encouraged to remain in the study until they have completed the 12 months follow-up. If the patient prematurely discontinues from the study, for any reason, a final evaluation must be completed for that patient and the reason for withdrawal must be documented. All documentation concerning the patients must be as complete as possible.

ELIGIBILITY:
I5.1 Inclusion criteria

* Patients must be previously diagnosed with type 2 diabetes with documented treatment with insulin, oral hypoglycemics, or diet controlled by medical history. (Undocumented or newly diagnosed diabetics must fulfill the American Diabetes Association Criteria-Report of the Expert Committee on the Diagnosis and Classification of Diabetes Mellitus (Diabetes Care 2003;26:S5-20)).
* Diagnosis of angina pectoris defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II-III) OR patients with documented silent ischemia;
* Patients with "de novo" coronary lesion (any length) who are eligible for coronary revascularization;
* Target lesion is ≥2.5 mm to ≤3.5mm in diameter (visual estimate);
* Target lesion stenosis is ≥50% (visual estimate);
* Male or Female age >18 years old;
* Patients with one or more lesions to be treated with a sirolimus eluting stent (Cypher, Cordis);
* Patient must provide written informed consent prior to the procedure using a form that is approved by the local Institutional Review Board.
* At least one lesion must be a complex lesion (see below for details)

5.2 Exclusion criteria

* Patients under age 18 years old;
* Patient has experienced an ST-segment elevation myocardial infarction within the preceding 30 days;
* Active liver disease (ALT>2.5 times upper limit of normal);
* Impaired renal function (creatinine ≥2.5 mg/dL);
* Previous brachytherapy of target vessel;
* Lesion of the Left Main trunk > 50%;
* Target lesion is in a saphenous venous graft or internal mammary graft;
* Target lesion is due to restenosis ;
* Recipient of heart transplant;
* Women who are pregnant or who have the potential to become pregnant during the study;
* Patients with life expectancy of less than one year or factors making clinical follow-up difficult;
* Patients with bleeding diathesis in whom anticoagulant or antiplatelet drug is contraindicated;
* Patient with intolerance/contraindication to Aspirin or Ticlopidine/Clopidogrel or pioglitazone treatment;
* Currently participating in an investigational drug or another device study;
* Patients with leukopenia;
* Patients with neutropenia;
* Documented peptic ulcer or gastric/intestinal bleeding in the last 6 months;
* Patients with thrombocytopenia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-12 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
In-Segment Late Loss | 9 months

SECONDARY OUTCOMES:
Binary restenosis | 9 months
MACE | 1, 9, 12 month
Stent thrombosis | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Romeo, MD, Study Chair — University of Rome Tor Vergata
Locations (1):
- Policlinico di Tor Vergata, Rome, Italy

REFERENCES:
- [Derived] Clementi F, Di Luozzo M, Mango R, Luciani G, Trivisonno A, Pizzuto F, Martuscelli E, Mehta JL, Romeo F. Regression and shift in composition of coronary atherosclerotic plaques by pioglitazone: insight from an intravascular ultrasound analysis. J Cardiovasc Med (Hagerstown). 2009 Mar;10(3):231-7. doi: 10.2459/JCM.0b013e3283212eb6. PMID 19262209
- See also: University web page — http://www.uniroma2.it
- See also: Hospital web page — http://www.ptvonline.it